CLINICAL TRIAL: NCT03828630
Title: Lung Ultrasound to Detect Pulmonary Complications in Critically Ill Parturients in an Urban Low-Resource Setting (LUSIP) - an Observational Study in Sierra Leone
Brief Title: Lung Ultrasound to Detect Pulmonary Complications in Critically Ill Parturients
Acronym: LUSIP
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Mahidol Oxford Tropical Medicine Research Unit (Other); University of Sierra Leone (Other); Doctors with Africa - CUAMM (Other); University of Bari (Other)
Responsible Party: Principal Investigator, Prof. Dr. Marcus J. Schultz, Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: LUSIP
Record Dates: First submitted 2019-01-29; First posted 2019-02-04 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Obstetric Complication; Lung Injury, Acute; Pulmonary Disease; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Acute Lung Injury; Lung Diseases; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims at describing the frequency, timing and type of pulmonary complications detected with lung ultrasound in critically-ill parturients in admitted to a high-dependency unit in Freetown, Sierra Leone.

DETAILED DESCRIPTION:
Rationale: The three big 'killers' in parturients, peripartum hemorrhage, sepsis and pre-eclampsia all predispose to pulmonary complications. These complications affect management before, during and after the primary obstetric problem has been solved. A timely diagnosis and thorough follow-up of pulmonary complications may benefit parturients. Lung ultrasound (LUS) is a point-of-care imaging bedside tool increasingly used in the critical care setting that may prove useful in parturients.

Objective: To describe frequency, timing and type of pulmonary complications detected with LUS in critically ill parturients in a high-dependency unit (HDU), and to determine the association with outcome.

Hypotheses: Pulmonary complications detected by LUS are frequent in parturients admitted to a HDU in a resource-limited setting, and are associated with hospital mortality.

Study design: A prospective observational study. Study population: Critically ill parturients admitted to the HDU of the Princess Christian Maternity Hospital (PCMH) in Freetown, Sierra Leone.

Sample size: No formal sample size calculation is performed. Based on current rates of admissions to the HDU of the PCMH the investigators expect to perform LUS in at least 125 patients.

Methods: A trained physician performs all 12-region LUS investigations. LUS is performed at admission, after 24 and 48 hours, and when a patient's respiratory condition deteriorates. LUS findings are reported using a standardized semi-quantitative visual LUS scoring method.

Main study parameters/primary endpoints: The proportion of critically ill parturients admitted to the HDU of the PCMH with pulmonary complications detected by LUS, including interstitial syndrome, pulmonary consolidation, and pleural effusion.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the HDU of the PCMH during the study period
* Verbal informed consent of the patient or his/her formal representative

Exclusion Criteria:

* Lung ultrasound not feasible, e.g., due to electricity breakdown, or absence of the trained sonographer.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Critically ill parturients admitted to the HDU of the Princess Christian Maternity Hospital (PCMH) in Freetown, Sierra Leone.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2018-07-08 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
Proportion of parturients with pulmonary complications | From admission to 48 hours later
  proportion of parturients with pulmonary complications detected by LUS during stay in the HDU.

SECONDARY OUTCOMES:
Description of lung ultrasound findings | From admission to 48 hours later
  Precise description of ultrasound findings (proportion of patients with a normal lung, interstitial syndrome, lung consolidation, pleural effusion)
Description of diagnoses made with lung ultrasound | From admission to 48 hours later
  Proportion of patients with a diagnosis of pneumonia, acute respiratory distress syndrome, fluid overload, no pulmonary complication.
Relative risk of death in patients with a pulmonary complication | On the day of HDU discharge or death, whichever came first, assessed up to 12 weeks after enrollment
  Risk of death in the group with pulmonary complication divided by the risk of death in parturients without a pulmonary complication

CONTACTS AND LOCATIONS:
Overall Officials: Marcella Schiavone, MD, PhD, Study Chair — Doctors with Africa - CUAMM; Anna de Nicolo, MD, PhD, Study Chair — University of Bari; Eva Henciles, MD, Principal Investigator — University of Sierra Leone; Marcus J Schultz, MD, PhD, Principal Investigator — University of Amsterdam
Locations (1):
- Princess Christian Maternity Hospital, Freetown, Sierra Leone

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Leopold SJ, Ghose A, Plewes KA, Mazumder S, Pisani L, Kingston HWF, Paul S, Barua A, Sattar MA, Huson MAM, Walden AP, Henwood PC, Riviello ED, Schultz MJ, Day NPJ, Kumar Dutta A, White NJ, Dondorp AM. Point-of-care lung ultrasound for the detection of pulmonary manifestations of malaria and sepsis: An observational study. PLoS One. 2018 Dec 12;13(12):e0204832. doi: 10.1371/journal.pone.0204832. eCollection 2018. PMID 30540757
- [Background] Vercesi V, Pisani L, van Tongeren PSI, Lagrand WK, Leopold SJ, Huson MMA, Henwood PC, Walden A, Smit M, Riviello ED, Pelosi P, Dondorp AM, Schultz MJ; Lung Ultrasound Consortium. External confirmation and exploration of the Kigali modification for diagnosing moderate or severe ARDS. Intensive Care Med. 2018 Apr;44(4):523-524. doi: 10.1007/s00134-018-5048-5. Epub 2018 Jan 24. No abstract available. PMID 29368056